CLINICAL TRIAL: NCT04137666
Title: NRS 2002: Nutritional Screen in Cancer Patients
Status: Completed | Type: Observational
Sponsor: Sociedad de Lucha Contra el Cáncer del Ecuador (Other)
Responsible Party: Sponsor
Other Study IDs: CISOLGYE20190020
Record Dates: First submitted 2019-10-22; First posted 2019-10-24 (Actual); Last update posted 2019-10-24 (Actual); Status verified 2019-10

CONDITIONS: Malnutrition (Diagnosis); Nutrition Disorders; Nutrition Surveys; Scoring System; Cancer; Nutrition Related Cancer
Keywords: Cancer Hospitalized Patients; Nutrition Disorders; Scoring System; Nutrition Surveys; Nutrition Assessment
MeSH Terms: conditions — Malnutrition; Disease; Nutrition Disorders; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Diagnosing the nutritional status of cancer patients is extremely important. An appropriate nutritional status supports a better tolerance to the treatment. A working protocol is essential to start with Nutritional Screening. If it is detected Malnutrition Risk or Malnutrition, diet counseling, and the specific therapeutic for each patient must be provided.

This descriptive study will serve three aims:

* Register in the cancer patient's electronic medical record their nutritional status at the admission and when the patient is discharged.
* Determine the percentage of malnourished patients or in the risk of malnutrition who are admitted to hospitalization.
* Recognize the number of patients that required specialized nutritional care.

The purpose of this study is to determine if 30% of the patients admitted to the headquarters of SOLCA in Guayaquil from the Ecuadorian Cancer Society are at malnutrition risk or with any specific malnutrition level.

DETAILED DESCRIPTION:
A prospective, descriptive, non-interventional study that will be performed from July 1st to October 4th of 2019 in all hospitalized patients of the Internal Medicine Service from SOLCA in Guayaquil from the Ecuadorian Cancer Society.

Statistical analysis: Central tendency measures. The results will be presented with tables and graphs.

Two weeks before the start of the study, the training of the personnel that will intervene in the screening of the participants will be carried out and will have a flow chart of actions to follow according to the status of patients.

ELIGIBILITY:
Inclusion Criteria:

* Participants older than 18-year old that go to the mentioned service

Exclusion Criteria:

* All patients with more than 48 hours of hospital admission
* Pediatric population.
* Patients with edema, non-malignant conditions (family of SOLCA workers) or with oncologic diagnosis not confirmed
* Participants who use a wheelchair or stretcher and those who cannot stand up

The NRS 2002 screening tool will be used to collect data and register the electronic medical record of each patient according to their nutritional status.

The variables to be recorded in an online Excel shared sheet (Google Drive) are weight, height, BMI, age, cancer diagnosis, associated comorbidities.

For weight determination, a scale (mechanical or electronic) in good condition will be used

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants older than 18-year old that go to the Internal Medicine Service from SOLCA in Guayaquil from the Ecuadorian Cancer Society, from July 1st to October 4th of 2019 in all hospitalized patients of
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Nutritional Status | 60 days
  Registration in the cancer patients' Clinical Record their nutritional status when they are admitted and when they are discharged
Percentage of malnourished patients or at risk of malnourishment | 60 days
  To know the percentage of malnourished patients or at risk of malnourishment that are admitted for hospitalization
Patients who needed specialized nutritional care | 60 days
  Recognize the number of patients who needed specialized nutritional care

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Oncológico Nacional Dr. Juan Tanca Marengo, Guayaquil, Guayas, Ecuador

REFERENCES:
- [Background] Pressoir M, Desne S, Berchery D, Rossignol G, Poiree B, Meslier M, Traversier S, Vittot M, Simon M, Gekiere JP, Meuric J, Serot F, Falewee MN, Rodrigues I, Senesse P, Vasson MP, Chelle F, Maget B, Antoun S, Bachmann P. Prevalence, risk factors and clinical implications of malnutrition in French Comprehensive Cancer Centres. Br J Cancer. 2010 Mar 16;102(6):966-71. doi: 10.1038/sj.bjc.6605578. Epub 2010 Feb 16. PMID 20160725
- [Background] Wie GA, Cho YA, Kim SY, Kim SM, Bae JM, Joung H. Prevalence and risk factors of malnutrition among cancer patients according to tumor location and stage in the National Cancer Center in Korea. Nutrition. 2010 Mar;26(3):263-8. doi: 10.1016/j.nut.2009.04.013. Epub 2009 Aug 8. PMID 19665873
- [Background] Rabito EI, Marcadenti A, da Silva Fink J, Figueira L, Silva FM. Nutritional Risk Screening 2002, Short Nutritional Assessment Questionnaire, Malnutrition Screening Tool, and Malnutrition Universal Screening Tool Are Good Predictors of Nutrition Risk in an Emergency Service. Nutr Clin Pract. 2017 Aug;32(4):526-532. doi: 10.1177/0884533617692527. Epub 2017 Feb 15. PMID 28199797
- [Background] Kondrup J, Rasmussen HH, Hamberg O, Stanga Z; Ad Hoc ESPEN Working Group. Nutritional risk screening (NRS 2002): a new method based on an analysis of controlled clinical trials. Clin Nutr. 2003 Jun;22(3):321-36. doi: 10.1016/s0261-5614(02)00214-5. PMID 12765673
- [Background] Cerezo, L. Diagnóstico del estado nutricional y su impacto en el tratamiento del cáncer. Oncolog. 2005; 28(3): 23-28.
- [Background] Gómez C, Rodríguez L, Luengo L, Zamora P, Celaya S, Zarazaga A. et al. Intervención nutricional en el paciente oncológico adulto. Barcelona: Glosa; 2003.
- [Background] Arends J, Bachmann P, Baracos V, Barthelemy N, Bertz H, Bozzetti F, Fearon K, Hutterer E, Isenring E, Kaasa S, Krznaric Z, Laird B, Larsson M, Laviano A, Muhlebach S, Muscaritoli M, Oldervoll L, Ravasco P, Solheim T, Strasser F, de van der Schueren M, Preiser JC. ESPEN guidelines on nutrition in cancer patients. Clin Nutr. 2017 Feb;36(1):11-48. doi: 10.1016/j.clnu.2016.07.015. Epub 2016 Aug 6. PMID 27637832
- [Background] Marin Caro MM, Gomez Candela C, Castillo Rabaneda R, Lourenco Nogueira T, Garcia Huerta M, Loria Kohen V, Villarino Sanz M, Zamora Aunon P, Luengo Perez L, Robledo Saenz P, Lopez-Portabella C, Zarazaga Monzon A, Espinosa Rojas J, Nogues Boqueras R, Rodriguez Suarez L, Celaya Perez S, Pardo Masferrer J. [Nutritional risk evaluation and establishment of nutritional support in oncology patients according to the protocol of the Spanish Nutrition and Cancer Group]. Nutr Hosp. 2008 Sep-Oct;23(5):458-68. Spanish. PMID 19160896